CLINICAL TRIAL: NCT01388309
Title: DAS Evaluation of RA Activity in Patients Treated With Tocilizumab
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis Who Have an Inadequate Response to DMARDs
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25524
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate in clinical practice the change in Disease Activity Score (DAS28) in patients with rheumatoid arthritis and an inadequate response to DMARDs who are initiated on treatment with RoActemra/Actemra (tocilizumab). Data will be collected from eligible patients (on 8 mg/kg or 4 mg/kg intravenously every 4 weeks, with or without methotrexate) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe active rheumatoid arthritis
* Inadequate response or intolerance to previous therapy with one or more traditional DMARDs

Exclusion Criteria:

* Pregnant or lactating women
* Active infection
* Positive for hepatitis B, hepatitis C or HIV infection
* Concomitant anti-TNF drugs
* Contraindications to treatment with RoActemra/Actemra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis and an inadequate response to DMARDs who are initiated on treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Disease activity score (DAS28) | 12 months

SECONDARY OUTCOMES:
DAS 28 (subgroup on monotherapy) | 12 months
DAS 28 (subgroup on 4 mg/kg dose) | 12 months
Safety: Incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Piešťany